CLINICAL TRIAL: NCT06012552
Title: Randomized, Double-blind, Placebo-controlled Trial of the Efficacy and Safety of Tianeptine in the Treatment of Covid Fog Symptoms in Patients After COVID-19 With the Study of the Pathophysiology of the Phenomenon Using Positron Emission Tomography, Biochemical, Immunological and Electrophysiological Parameters.
Brief Title: Randomized, Double-blind, Placebo-controlled Trial of the Efficacy and Safety of Tianeptine in the Treatment of Covid Fog Symptoms in Patients After COVID-19.
Acronym: COVMENT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Collaborators: ABM Industries (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABM/COVMENT/2021; 2022-000893-25 (EudraCT Number)
Record Dates: First submitted 2023-08-24; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Nervous System Diseases
Keywords: COVID-19; memory problems; Covid Fog; brain fog; COVID-19 brain fog; lack of mental clarity; poor concentration; headaches; confusion
MeSH Terms: conditions — Nervous System Diseases; COVID-19; Memory Disorders; Mental Fatigue; Headache; Confusion | interventions — tianeptine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stady group (Experimental): The study group will receive oral tianeptine in a dose of 3x 12.5 mg per day (patients younger than 70) or 2x 12.5 mg per day (patients older than 70) for 16 weeks. In addition, the subjects will participate in group psychotherapy and neurological rehabilitation.
  Interventions: Drug: Tianeptine
- Control group (Placebo Comparator): The control group will receive oral placebo in a dose of 3x 12.5 mg per day (patients younger than 70) or 2x 12.5 mg per day (patients older than 70) for 16 weeks. In addition, the subjects will participate in group psychotherapy and neurological rehabilitation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tianeptine — Tianesal 12,5mg
  Arms: Stady group
Drug: Placebo — application as in the control group
  Arms: Control group

SUMMARY:
COVID-19 is associated with a high risk of complications from the central nervous system. Syndrome of cognitive disorders- in terms of memory, attention or executive functions among COVID-19 convalescents is often called brain fog (covid fog - CF). CF leads to psychomotor retardation and chronic fatigue syndrome, resulting in poor functioning and low quality of life. CF may affect up to 81% of patients after COVID-19.

Prevalence of CF may be even greater among patients with severe forms of COVID-19. In the preliminary assessment authors found that 83% of COVID-19 inpatients had at least mild cognitive impairment. Moreover, SARS-CoV-2 infection is associated with higher incidence of depression and anxiety disorders. CF pathogenesis is not fully understood. There exist no strict diagnostic criteria for it, as well as no therapeutic recommendations. Health care systems of many countries, including Poland, lack therapeutic programs addressed at patients with CF. Tianeptine may be a drug with potentially beneficial effects in CF. Neuroprotective, antidepressive, sleep-improving and anxiolytic properties of tianeptine allow it to choose as a candidate for CF amelioration. There is also data supporting the thesis that patients with CF may benefit from short-term group therapy. It has been proven to improve quality of life, reduce stress, and improve cognitive function in non-MC cognitive disorders.

Expected research results: A database will be created from the collected clinical, laboratory and additional data. Statistical models will be created to predict: the duration of disorders, response to therapy, the final result of treatment. Among the markers of CNS damage, those which correlates with the patient's condition will be selected.

The study will allow to estimate the prevalence of CF in the population. PET-CT and auditory evoked potentials also will be used to expand knowledge in the field of CF.

Based on the existing data, an improvement is expected in all investigated participants as a result of rehabilitation and psychotherapy.

Additional improvement is expected in the tianeptine group. Improvement will be defined as: reduction in the severity of anxiety and depression disorders, reduction in the severity of cognitive disorders, improvement in the quality of life. The results will be used to develop a new diagnostic and therapeutic pathway and a comprehensive intervention program in CF.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient to participate in the clinical trial.
* Age ≥ 18 years.
* History of COVID-19 infection confirmed by a positive SARS-CoV-2 test result by RT- PCR or positive antigen test.
* Subjective patient-reported cognitive decline after COVID-19 infection at Screening.
* Cognitive dysfunction found at Screening, defined by the Montreal Scale for the Assessment of Cognitive Function (MoCA) as a score of less than 26.
* Use of effective contraception by women of childbearing potential.

Exclusion Criteria:

* Hypersensitivity to tianeptine.
* Hypersensitivity to fluorodesoxyglucose (FDG).
* History of allergy to drugs or other substances, which, in the Investigator's opinion, is a contraindication to participation in the study.
* History of stroke.
* Ever undergone and planned brain surgery at the time of the study.
* Previously diagnosed organic damage to the central nervous system.
* Diagnosed organic mental disorder.
* Diagnosed bipolar affective disorder.
* Diagnosed psychotic disorder.
* History of active depressive episode, including those diagnosed at the time of study eligibility, requiring antidepressant treatment.
* Diagnosed mental retardation.
* Bipolar affective disorder in a first-degree relative.
* Uncontrolled diabetes mellitus.
* Severe renal failure with eGFR < 30ml/min/1.73 m2.
* cirrhosis of liver Severe liver cirrhosis (Child-Pugh class C ).
* Claustrophobia.
* Diagnosed chronic diseases that significantly worsen the patient's prognosis and quality of life, which, in the Investigator's opinion, may adversely affect the patient's participation in the study.
* Active or past malignancy within the past 5 years, except for basal cell carcinoma of the skin and cervical cancer in situ in patients who have received radical treatment.
* Active viral, bacterial, fungal, tuberculous, or parasitic infection.
* History or presence of other relevant diseases which, in the Investigator's opinion, is a contraindication to participation in the study.
* Positive pregnancy test performed on women of childbearing potential at screening or Visit 1.
* Taking medications:

  1. Non-selective MAO inhibitors within 14 days prior to screening,
  2. Mianserin during screening.
* Significant difficulty with peripheral venous cannulation.
* Positive history of alcohol, drug, and psychoactive abuse/dependence.
* Pregnancy or planning a pregnancy during the study period.
* Breastfeeding or planning to breastfeed during the study period.
* Current participation in another clinical trial.
* Lack of patient compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in covid fog symptoms | 16 week after randomization
  Improvement in covid fog symptoms at week 16 after randomization defined as a 2 point improvement in MoCA score.

SECONDARY OUTCOMES:
improving cognitive function | 16 week after randomization
  Complete resolution of covid fog symptoms at week 16 after randomization defined as normalization of MoCA scale score (MoCA = 26
  - 30 points).
Change in brain metabolic activity | 16 week after randomization
  Change in brain metabolic activity as assessed by PET-CT at week 16 after randomization.

CONTACTS AND LOCATIONS:
Locations (1):
- Anna Klimkiewicz, Warsaw, Poland